CLINICAL TRIAL: NCT05314231
Title: A Phase 1b, Open-Label, Single-Dose Pharmacokinetic Study of Subcutaneous ALXN1720 in Adult Participants With Varying Degrees of Proteinuria
Brief Title: Safety and Pharmacokinetic Study of Subcutaneous ALXN1720 in Participants With Proteinuria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1720-NEPH-102
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Proteinuria
Keywords: Proteinuria; Glomerular Disease; Chronic Kidney Disease; Lupus Nephritis; Immunoglobulin A Nephropathy; Primary Membranous Nephropathy; Focal Segmental Glomerulosclerosis; Diabetic Nephropathy; Hypertensive Nephrosclerosis; Minimal Change Disease; Thin Basement Membrane Nephropathy; Membranoproliferative Glomerulonephritis (all forms)
MeSH Terms: conditions — Proteinuria; Renal Insufficiency, Chronic; Lupus Nephritis; Glomerulonephritis, IGA; Glomerulosclerosis, Focal Segmental; Diabetic Nephropathies; Nephrosis, Lipoid; Hematuria, Benign Familial; Glomerulonephritis, Membranoproliferative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALXN1720 (Experimental): Participants will receive a single dose of ALXN1720, given as a SC infusion at a dose of 1500 mg.
  Interventions: Drug: ALXN1720

INTERVENTIONS:
Drug: ALXN1720 — All enrolled participants will receive a single dose of ALXN1720 on Day 1 followed by a Post-treatment and Follow-up Period (92 days).

SUMMARY:
The primary objective of this study is to assess the impact of proteinuria on the pharmacokinetic (PK) of a single dose of ALXN1720 in participants with proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Lupus Nephritis, IgA Nephropathy, Primary Membranous Nephropathy, Focal Segmental Glomerulosclerosis, Diabetic Nephropathy, Hypertensive Nephrosclerosis, Minimal Change Disease, Thin Basement Membrane Nephropathy or Membranoproliferative Glomerulonephritis (all forms). Other cause of kidney disease may be included per investigator agreement with the Sponsor
* Proteinuria >=1 based on absolute amount in grams per day (g/d) as measured in one complete and valid 24-hour urine collection during Screening
* Body weight ≥ 40 kg at Screening

Exclusion Criteria:

* Kidney transplant
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 during Screening
* Known medical or psychological condition(s) or risk factor that, in the opinion of the Investigator, might interfere with the participant's full participation in the study, pose any additional risk for the participant, or confound the assessment of the participant or outcome of the study.
* Treatment with complement inhibitors at any time.
* Treatment with rituximab within 6 months before initiation of study drug on Day 1; or, planned treatment with rituximab within 3 months after initiation of study drug on Day 1.
* Participation in another investigational drug or investigational device study within 30 days before initiation of study drug on Day 1 in this study or within 5 half-lives of that investigational product, whichever is greater.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Serum Concentration of ALXN1720 | Day 1 (0.5 hours predose and postdose) and postdose on Days 2, 3, 8, 15, 29, 43, and 57

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events | Day 1 (Predose) through Follow-up (Day 92)
Serum Concentration of Free and Total Complement Component 5 (C5) | Day 1 (0.5 hours predose and postdose) and postdose on Days 2, 3, 8, 15, 29, 43, and 57
Number of Participants With Antidrug Antibodies (ADAs) to ALXN1720 | Day 1 (predose) through Day 57

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Clinical Trial Site 2, Anyang-si, Gyeonggi-do
  - Clinical Trial Site 1, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.